CLINICAL TRIAL: NCT03000075
Title: A Phase II/III, Randomized, Double-blind Study to Evaluate Efficacy and Safety of Two Different Dose Regimens of BI 655066 (Risankizumab) and Placebo and Maintenance of Response of BI 655066 (Risankizumab) Administered Subcutaneously in Japanese Patients With Moderate to Severe Chronic Plaque Type Psoriasis.
Brief Title: BI 655066 (Risankizumab) Compared to Placebo in Japanese Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M16-004; 1311.38 (Other: Boehringer Ingelheim)
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Psoriasis
Keywords: BI 655066; ABBV-066; risankizumab
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Part A) (Placebo Comparator): Participants randomized to receive double-blind (DB) placebo for risankizumab by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: placebo for risankizumab
- Risankizumab 75 mg (Part A) (Experimental): Participants randomized to receive double-blind (DB) risankizumab 75 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: risankizumab; Drug: placebo for risankizumab
- Risankizumab 150 mg (Part A) (Experimental): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — Risankizumab pre-filled syringe, administered by subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066
  Arms: Risankizumab 150 mg (Part A); Risankizumab 75 mg (Part A)
Drug: placebo for risankizumab — Placebo for risankizumab pre-filled syringe, administered by subcutaneous (SC) injection
  Arms: Placebo (Part A); Risankizumab 75 mg (Part A)

SUMMARY:
This is a randomized double blind, double dummy, placebo controlled, parallel design study that is being performed to assess the safety and efficacy of BI 655066 (risankizumab).

DETAILED DESCRIPTION:
Participants were randomized to receive either placebo, risankizumab 75 mg, or risankizumab 150 mg in Part A. All participants received 2 injections to maintain the blind: the placebo arm received 2 injections of placebo, the risankizumab 75 mg arm received one injection of risankizumab 75 mg and one injection of placebo, and the risankizumab 150 mg arm received 2 injections of risankizumab 75 mg. Participants who received placebo in Part A switched to risankizumab in Part B; participants who received risankizumab (75 mg or 150 mg) in Part A continued to receive the same treatment (risankizumab 75 mg or 150 mg) in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of chronic plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before the first administration of study drug. Duration of diagnosis may be reported by the patient.
* Have stable moderate to severe chronic plaque psoriasis with or without psoriatic arthritis at both Screening and Baseline (Randomisation):

  1. Have an involved body surface area (BSA) ≥10% and
  2. Have a Psoriasis Area and Severity Index (PASI) score ≥12 and
  3. Have a Static Physician Global Assessment (sPGA) score of ≥3.

Exclusion Criteria:

* Patients with

  1. non-plaque forms of psoriasis (including guttate, erythrodermic, or pustular)
  2. current drug-induced psoriasis (including an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
  3. active ongoing inflammatory diseases other than psoriasis and psoriatic arthritis that might confound trial evaluations according to investigator's judgment
* Previous exposure to BI 655066

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2018-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

REFERENCES:
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- [Derived] Ohtsuki M, Fujita H, Watanabe M, Suzaki K, Flack M, Huang X, Kitamura S, Valdes J, Igarashi A. Efficacy and safety of risankizumab in Japanese patients with moderate to severe plaque psoriasis: Results from the SustaIMM phase 2/3 trial. J Dermatol. 2019 Aug;46(8):686-694. doi: 10.1111/1346-8138.14941. Epub 2019 Jun 25. PMID 31237727

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 182 subjects were enrolled; 11 subjects failed screening and are excluded from the analyses.
Groups:
- Placebo/Risankizumab 75 mg (Part B): Participants randomized to receive placebo in Part A switched to risankizumab 75 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Placebo/Risankizumab 150 mg (Part B): Participants randomized to receive placebo in Part A switched to risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Risankizumab 75 mg/Risankizumab 75 mg (Part B): Participants randomized to receive risankizumab 75 mg in Part A continued to receive risankizumab 75 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
- Risankizumab150 mg /Risankizumab 150 mg (Part B): Participants randomized to receive risankizumab 150 mg in Part A continued to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
Period: Part A
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A) | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Started | 58 | 58 | 55 | 0 | 0 | 0 | 0
Completed | 54 | 58 | 55 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A) | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Started | 0 | 0 | 0 | 27 (Participants who received placebo in Part A received risankizumab 75 mg in Part B) | 27 (Participants who received placebo in Part A received risankizumab 150 mg in Part B) | 58 (Participants who received risankizumab 75 mg in Part A received risankizumab 75 mg in Part B) | 55 (Participants who received risankizumab 150 mg in Part A received risankizumab 150 mg in Part B)
Completed | 0 | 0 | 0 | 27 | 26 | 56 | 54
Not Completed | 0 | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Not dosed due to AE | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A) | Total
Number analyzed (Participants) | 58 | 58 | 55 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.24) | 51.5 (12.33) | 53.3 (11.94) | 51.9 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 5 | 28
  Male | 45 | 48 | 50 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 58 | 58 | 55 | 171
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 58 | 58 | 55 | 171
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: Intent-to-treat (ITT) population: all participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A)
Number analyzed (Participants) | 58 | 58 | 55
percentage of participants | 1.7 | 75.9 | 74.5
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab 75 mg (Part A); Test type: Other — Cochran-Mantel-Haenszel test adjusted for strata: weight (≤ 90 kg vs > 90 kg) and concomitant psoriatic arthritis (PsA) at Baseline (YES: DIAGNOSED or SUSPECTED vs NO). If there was a stratum containing zero count, 0.1 was added to each cell; p < 0.001, Cochran-Mantel-Haenszel — P-value was calculated from the Cochran-Mantel-Haenszel test adjusted for strata. If there was a stratum containing zero count, 0.1 was added to each cell; Adjusted percentage difference = 73.6, 95% CI 2-sided [62.2 to 85.0] — 95% confidence interval (CI) for adjusted difference of 2 treatment groups, calculated from the Cochran-Mantel-Haenszel test adjusted for strata. If there was a stratum containing zero count, 0.1 was added to each cell
Statistical Analysis 2: Comparison: Placebo (Part A) vs Risankizumab 150 mg (Part A); Test type: Other — Cochran-Mantel-Haenszel test adjusted for strata: weight (≤ 90 kg vs > 90 kg) and concomitant PsA at Baseline (YES: DIAGNOSED or SUSPECTED vs NO). If there was a stratum containing zero count, 0.1 was added to each cell; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 72.4, 95% CI 2-sided [60.6 to 84.1] — 95% CI for adjusted difference of 2 treatment groups, calculated from the Cochran-Mantel-Haenszel test adjusted for strata. If there was a stratum containing zero count, 0.1 was added to each cell

2. Secondary Outcome: Percentage of Participants Achieving PASI90 at Week 52 (Part B)
Description: as for outcome 1
Time Frame: Week 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Number analyzed (Participants) | 27 | 27 | 58 | 55
percentage of participants | 81.5 | 85.2 | 86.2 | 92.7

3. Secondary Outcome: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of Clear or Almost Clear at Week 16 (Part A)
Description: The sPGA is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA ranges from 0 to 4, and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A)
Number analyzed (Participants) | 58 | 58 | 55
percentage of participants | 10.3 | 86.2 | 92.7
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab 75 mg (Part A); Cochran-Mantel-Haenszel test adjusted for strata: weight (≤ 90 kg vs > 90 kg) and concomitant PsA at Baseline (YES: DIAGNOSED or SUSPECTED vs NO). If there was a stratum containing zero count, 0.1 was added to each cell; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 75.0, 95% CI 2-sided [63.8 to 86.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo (Part A) vs Risankizumab 150 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 82.4, 95% CI 2-sided [72.2 to 92.6] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants Achieving sPGA Score of Clear or Almost Clear at Week 52 (Part B)
Description: as for outcome 3
Time Frame: Week 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Number analyzed (Participants) | 27 | 27 | 58 | 55
percentage of participants | 96.3 | 88.9 | 84.5 | 94.5

5. Secondary Outcome: Percentage of Participants Achieving 75% Improvement in PASI Score (PASI75) at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI75 is defined as at least a 75% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A)
Number analyzed (Participants) | 58 | 58 | 55
percentage of participants | 8.6 | 89.7 | 94.5
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab 75 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 80.3, 95% CI 2-sided [70.1 to 90.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo (Part A) vs Risankizumab 150 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 86.0, 95% CI 2-sided [76.8 to 95.1] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Percentage of Participants Achieving PASI75 at Week 52 (Part B)
Description: as for outcome 5
Time Frame: Week 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Number analyzed (Participants) | 27 | 27 | 58 | 55
percentage of participants | 100 | 88.9 | 94.8 | 96.4

7. Secondary Outcome: Percentage of Participants Achieving 100% Improvement in PASI Score (PASI100) at Week 16 (Part A)
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI100 is defined as a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A)
Number analyzed (Participants) | 58 | 58 | 55
percentage of participants | 0 | 22.4 | 32.7
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab 75 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 22.6, 95% CI 2-sided [11.8 to 33.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo (Part A) vs Risankizumab 150 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 32.5, 95% CI 2-sided [20.0 to 45.0] — [estimate comment as in outcome 1, analysis 2]

8. Secondary Outcome: Percentage of Participants Achieving PASI100 at Week 52 (Part B)
Description: as for outcome 7
Time Frame: Week 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Number analyzed (Participants) | 27 | 27 | 58 | 55
percentage of participants | 40.7 | 44.4 | 43.1 | 41.8

9. Secondary Outcome: Percentage of Participants (ITT Participants in Select Study Sites With Confirmed Diagnosis of Psoriatic Arthritis and Baseline Total Tender and Swollen Joint Count ≥ 3) Achieving an American College of Rheumatology 20 Response (ACR20) at Week 16 (Part A)
Description: Response defined by ACR20 criteria (improvement from baseline): ≥ 20% improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of the 5 following parameters: Patient assessment of pain; Patient global assessment of disease activity; Investigator's global assessment of disease activity; Health Assessment Questionnaire Disability Index (HAQ-DI); and Acute phase reactant value (C-reactive protein). Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Population: Among participants with confirmed diagnosis of PsA using classification criteria for psoriatic arthritis (CASPAR) and with baseline total tender joint count (TJC) and swollen joint count (SJC) counts ≥ 3 at selected study sites of the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A)
Number analyzed (Participants) | 3 | 5 | 3
percentage of participants | 0 | 40.0 | 33.3
Statistical Analysis 1: Comparison: Placebo (Part A) vs Risankizumab 75 mg (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Other; p = 0.131, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 39.2, 95% CI 2-sided [-11.6 to 90.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo (Part A) vs Risankizumab 150 mg (Part A); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.269, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Adjusted percentage difference = 31.3, 95% CI 2-sided [-24.2 to 86.7] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Percentage of Participants (ITT Participants in Select Study Sites With Confirmed Diagnosis of Psoriatic Arthritis and Baseline Total Tender and Swollen Joint Count ≥ 3) Achieving an ACR20 at Week 52 (Part B)
Description: as for outcome 9
Time Frame: Week 52
Population: Among participants with confirmed diagnosis of PsA using CASPAR criteria and with baseline TJC and SJC counts ≥ 3 at selected study sites of the ITT population,
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab150 mg /Risankizumab 150 mg (Part B)
Number analyzed (Participants) | 1 | 2 | 5 | 3
percentage of participants | 100 | 100 | 60.0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 16 weeks after the last dose of study drug (up to 56 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 16 weeks after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Risankizumab 150 mg (Part A): ): Participants randomized to receive double-blind (DB) risankizumab 150 mg by subcutaneous (SC) injection at Weeks 0 and 4 (Part A).
- Risankizumab 150 mg/Risankizumab 150 mg (Part B): Participants randomized to receive risankizumab 150 mg in Part A continued to receive risankizumab 150 mg by subcutaneous (SC) injection at Weeks 16, 28, and 40 (Part B).
Arm/Group | Placebo (Part A) | Risankizumab 75 mg (Part A) | Risankizumab 150 mg (Part A) | Placebo/Risankizumab 75 mg (Part B) | Placebo/Risankizumab 150 mg (Part B) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) | Risankizumab 150 mg/Risankizumab 150 mg (Part B)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/55 | 0/27 | 0/27 | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 1/58 | 2/58 | 2/55 | 2/27 | 0/27 | 1/56 | 1/54
Other Adverse Events (participants affected / at risk) | 22/58 | 14/58 | 14/55 | 10/27 | 19/27 | 23/56 | 19/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=58) | Risankizumab 75 mg (Part A) (N=58) | Risankizumab 150 mg (Part A) (N=55) | Placebo/Risankizumab 75 mg (Part B) (N=27) | Placebo/Risankizumab 150 mg (Part B) (N=27) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) (N=56) | Risankizumab 150 mg/Risankizumab 150 mg (Part B) (N=54)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Part A) (N=58) | Risankizumab 75 mg (Part A) (N=58) | Risankizumab 150 mg (Part A) (N=55) | Placebo/Risankizumab 75 mg (Part B) (N=27) | Placebo/Risankizumab 150 mg (Part B) (N=27) | Risankizumab 75 mg/Risankizumab 75 mg (Part B) (N=56) | Risankizumab 150 mg/Risankizumab 150 mg (Part B) (N=54)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 8 (8) | 3 (4) | 10 (11) | 8 (8) | 8 (12) | 12 (13) | 11 (12)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-06-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03000075/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03000075/SAP_003.pdf